CLINICAL TRIAL: NCT04803136
Title: The Role of Bone SPECT/CT in Evaluation of Persistent or Recurrent Back Pain Following Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Raghda Hassan Mohamed Farweiz, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SPECT/CT after spine surgery
Record Dates: First submitted 2021-01-19; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Spine Fusion
Keywords: Bone SPECT/CT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone SPECT/CT (Other): Gamma Camera with computed tomography
  Interventions: Procedure: spine surgeries
- Spine surgeries (Other): spine stabilization and fusion surgeries
  Interventions: Procedure: spine surgeries

INTERVENTIONS:
Procedure: spine surgeries — all spine surgeries including stabilization and fusion surgeries

SUMMARY:
* To evaluate the role of SPECT/CT in assessment of the osteoblastic activity in patients with persistent or recurrent back pain after spine surgery with inconclusive CT/MRI findings.
* To assess the value of bone SPECT/CT in the management of back pain.

DETAILED DESCRIPTION:
Low back pain is a common disorder, with international studies having found prevalence rates between 12% and 35% and life time prevalence rates ranging from 49% to 80%.

It is caused mainly by degenerative spinal disorders, such as spondylolisthesis, degenerative scoliosis, degenerative disc disease and recurrent disc herniations.

The management of low back pain varies from conservative to more invasive methods, such as spinal stabilization surgery that involves the placement of metallic screws, rods, plates or cages. Such surgery is increasingly performed to improve spinal stability in a variety of spine pathologies, including disc degeneration, spinal stenosis and spondylolisthesis.

On the other hand, spinal fusion surgery is performed in patients with severe chronic back pain when segmental instability is believed to cause the symptoms. The rationale for this is that pain relief will be achieved once the fusion restricts motion in the painful segments. For this purpose, a wide array of techniques has been proposed, including dorsal or dorsoventral spondylodesis, either in a one-step or two-step procedure.

It is estimated that more than 300,000 lumbar spinal fusion procedures are performed annually in the United States, and a continuously rising trend has also been observed in other parts of the world.

Unfortunately, recurrent pain after spinal surgery is a well known problem. It is reported that up to 10-20% of patients experience persistent/recurrent pain after lumbar spinal instrumentation and fusion , with studies estimating the surgical reintervention rate to be around 14% over a 4-year follow-up period and 19% over 11 years.

This may be related to loosening of the metallic implants or to a failure of a stably implanted graft to immobilize the fused segments. A further differential diagnosis is degenerative disease involving the spinal segments above or below the instrumented region. This so-called adjacent instability (AI) or adjacent level disease (ALD) may be precipitated by arthrodesis, as this procedure alters the biomechanics of the spine, thereby increasing motion of a mechanical load on the segments neighboring the graft. The differentiation between these conditions has therapeutic consequences as the treatment varies according to the cause.

Standard evaluation of patients with persistent or recurrent pain following spinal stabilization surgery includes clinical examination and conventional imaging using plain radiography, CT or MR imaging.

Conventional imaging is performed for the evaluation of hardware position (changes), hardware failure, fusion evolution, alignment of the vertebrae, possible pseudarthrosis and hardware loosening.

In general, because of the presence of nonspecific postoperative changes and metal-related imaging artifacts, the interpretation of CT images is often challenging and inconclusive. Thus, whether surgical reintervention is indicated based on conventional imaging may prove difficult to ascertain.

The value of bone scintigraphy with single-photon emission tomography/computed tomography (SPECT/CT) in patients with persistent or recurrent back pain after spine stabilization surgery has been addressed in a number of studies and the technique has been suggested to be a useful diagnostic tool for identification of postsurgical spine pathology.

Although most of these studies were based on a small sample size and lacked robust reference standards; it has been concluded that the use of SPECT/CT adds value in assessing patients following spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent/recurrent back pain after spine surgery and inconclusive conventional imaging.
* All patients will be clinically assessed by orthopedic surgeons or neurosurgeons specialized and experienced in spine surgery.

Exclusion Criteria:

* Patients less than 18 years old.
* Patients in whom stabilization surgery is secondary to a destructive bone malignancy (including multiple myeloma).
* Patients with known metabolic bone disease (such as Rheumatoid Arthritis, AS & SLE)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
use of SPECT/CT to measure the level of pain either persistent or recurrent after spine stabilization and fusion surgeries at any level of the spine and give a score and make a pain scale before and after therapeutic injection | up to 2 years
  Patients complaining from persistent or recurrent pain after spine stabilization and fusion surgeries at any level of the spine up to two years after surgery do CT/MRI and give inconclusive results, those patients referred to do Single Photon Emission Tomography/Computed Tomography at nuclear medicine unit using radioactive material Technicium99m- Methylene Diphosphonate to measure any increase in osteoblastic activity in the region of the stabilized segment for example at adjacent facet joint, sacrum or endplates and compare it with iliac crest activity then give therapeutic injection at determined increased activity and make pain score before and after therapeutic injection then follow up after 15 days

REFERENCES:
- [Background] Taylor J. Imaging in radiotherapy: looking to the future. Radiogr Today. 1989 Jul;55(626):16-9. No abstract available. PMID 2686691
- [Background] Mathew B, Norris D, Mackintosh I, Waddell G. Artificial intelligence in the prediction of operative findings in low back surgery. Br J Neurosurg. 1989;3(2):161-70. doi: 10.3109/02688698909002791. PMID 2679685
- [Background] Holch M, Grob PJ, Fierz W, Glinz W, Geroulanos S. [Immunosuppression caused by surgery and severe trauma]. Helv Chir Acta. 1989 Jun;56(1-2):121-4. German. PMID 2777589
- [Background] Fisher MA. SSEP in lumbar radiculopathy. Neurology. 1990 Feb;40(2):386-7. doi: 10.1212/wnl.40.2.386-a. No abstract available. PMID 2153944